CLINICAL TRIAL: NCT07251504
Title: Mitochondrial Metabolism and Oxidative Stress in Function of the Type of Physical Exercise and Nutritional Counseling in Type 2 Diabetes Mellitus
Brief Title: Mitochondrial Metabolism and Oxidative Stress in Function of the Physical Exercise and Nutritional Counseling in T2DM
Acronym: MITOX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MITOX; PP11-007-2023 (Other Grant/Funding Number: Instituto de Investigación e Innovación Biomédica de Cádiz)
Record Dates: First submitted 2025-09-26; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: metabolic disorders; aerobic exercise; muscle metabolism; high-resolution respirometry
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: The project is a randomized controlled trial in individuals with type 2 diabetes and obesity
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ND-INACT (No Intervention): Participants who did not receive either nutritional intervention or exercise program. They were instructed to maintain their normal life habits regarding physical activity and diet.
- Moderate-intensity continuous training (ND-MICT) (Active Comparator): Participants who did not receive nutritional intervention but were enrolled in a moderate-intensity continuous training exercise program.
  Interventions: Other: The Moderate-Intensity Continuous Training (MICT)
- High-intensity interval training (ND-HIIT) (Active Comparator): Participants who did not receive nutritional intervention but were enrolled in a high-intensity interval training exercise program.
  Interventions: Other: The High-Intensity Interval Training (HIIT)
- Nutritional intervention (D-INACT) (Active Comparator): Participants who received nutritional intervention but not an exercise program.
  Interventions: Behavioral: Nutritional intervention
- Nutritional Intervention Moderate-Intensity continuous training (D-MICT) (Experimental): Participants who received nutritional intervention and were enrolled in a moderate-intensity continuous training exercise program.
  Interventions: Behavioral: Nutritional intervention; Other: The Moderate-Intensity Continuous Training (MICT)
- Nutritional Intervention High-intensity interval training (D-HIIT) (Experimental): Participants who received nutritional intervention and were enrolled in a high-intensity interval training exercise program.
  Interventions: Behavioral: Nutritional intervention; Other: The High-Intensity Interval Training (HIIT)

INTERVENTIONS:
Behavioral: Nutritional intervention — The nutritional intervention was conducted through biweekly (± 3 days) in-person consultations with a nutritionist or dietitian over an entire period of 12 weeks. Firstly, the patient's diet was analyzed. Then, participants were guided to follow a Mediterranean pattern-based and mildly calorie-restricted diet, with the primary goal of achieving a 5 % reduction in body weight and reducing blood glucose levels. Meal plans were created using Nutrium® software , personalized to each participant's lifestyle and food preferences, and reviewed at each biweekly consultation. The dietary plan included at least 4 meals per day, ensuring a well-distributed intake of carbohydrates, a balanced distribution of macro- and micronutrients, and the inclusion of foods rich in prebiotics and probiotics. Moreover, some suggestions about the combination of foods and culinary techniques were provided. Only one session through the intervention was allowed to be attended telephonically.
  Arms: Nutritional Intervention High-intensity interval training (D-HIIT); Nutritional Intervention Moderate-Intensity continuous training (D-MICT); Nutritional intervention (D-INACT)
Other: The High-Intensity Interval Training (HIIT) — Participants assigned to the HIIT completed 3 weekly sessions, with 1-2 days of rest between sessions, on a cycle ergometer for 12 weeks.
  The training load (TL) was determined from an incremental test until volitional exhaustion with one-minute work intervals (from 85% to 165% of maximal power output from a previously performed VO2max test [Wmax] and with 10% increments) separated by 1.5-minute rest periods (at 20% Wmax).
  The program consisted of a 3 minutes warm-up with the first 2 minutes at 20% and last minute at 40% of the TL, followed by 10 series of 1 min duration at 90% of TL, with 1 minute of rest between sets at 40% of TL and ending with 2 minutes of cool-down at 20% of TL (estimated total time of the session: 25 minutes). A 5% increase in workload was applied when, for two consecutive sessions, the first three intervals failed to exceed 85%, and the last five did not reach 90% of maximal HR. Participants were asked to maintain a cadence above 80RPM.
  Arms: High-intensity interval training (ND-HIIT); Nutritional Intervention High-intensity interval training (D-HIIT)
Other: The Moderate-Intensity Continuous Training (MICT) — Participants assigned to the MICT completed 3 weekly sessions, with 1-2 days of rest between sessions, on a cycle ergometer for 12 weeks.
  MICT consisted of 50 minutes of continuous pedaling at an intensity approximately 10 % above the lactate threshold, with a cadence between 60-80 rpm. Training load (TL) was increased by 10% if these two conditions were met: 1) no increase of at least 2 beats of heart rate from minute 20 to minute 40 of the training session, and 2) lactate levels below 2 mmol/L in minute 48 of the session. The TL for the first session was determined by an adjustment test consisting of an incremental test with five consecutive 10-minute phases at a constant cadence (60-80 RPM) from 90% to 130% of the ventilatory threshold power, calculated from previously performed FatOx test data, with 10% increments in each step. TL was determined by the phase in which HR increased by ≥ 3 beats between phases and blood lactate levels increased by ≥ 1 mmol/L from the previous phase.
  Arms: Moderate-intensity continuous training (ND-MICT); Nutritional Intervention Moderate-Intensity continuous training (D-MICT)

SUMMARY:
The goal of this randomized controlled trial is to learn about the effects of different aerobic modalities (moderate-intensity continuous training (MICT) and high-intensity interval training (HIIT)) and diet on mitochondrial properties and oxidative stress in patients with type 2 diabetes (T2D). It will also learn about the different effects of these interventions in men and women. The main questions it aims to answer are:

* What is the isolated and combined effect of these exercise modalities and diet? Is there a superior approach for mitochondrial metabolism and oxidative stress in patients with T2D?
* Is there a sex-specific best combination choice for these different interventions?
* Is there any relation between exercise and diet-induced changes in mitochondrial properties and oxidative stress and other health-related outcomes such as body composition or insulin sensitivity?

To answer these questions, researchers designed a two-factor study. One factor was exercise, which had three levels (MICT, HIIT, and the inactive (INACT) condition). The second factor was diet, with two levels (Diet (D) and no diet (ND)). Hence, participants were randomly allocated into 6 groups: INACT-ND, INACT-D, MICT-ND, MICT-D, HIIT-ND, and HIIT-D.

Participants did:

* Underwent a 12-week intervention within the condition of his/her group
* Visit the research group facilities three times per week if in an exercise group or once every two weeks if in a diet group.

DETAILED DESCRIPTION:
This is a randomized controlled trial conducted in the Province of Cádiz (Spain). A total of 146 participants were enrolled in the study and underwent baseline and post-intervention determinations of the study outcomes. Just after the baseline determination, participants were randomly allocated to one of the aforementioned study groups. The randomization process was stratified by sex, which means that approximately 50% of participants in each group were women. All participants received detailed written and verbal information about the study objectives, procedures, benefits, and potential risks before providing written informed consent. This study adhered to the principles of the Declaration of Helsinki and was approved by the Provincial Research Ethics Committee of Cádiz and the Coordinating Committee of Biomedical Research Ethics of Andalucía (registration number 92.21; PEIBA number 1026-N-21; internal codes SICEIA-2025-001870 and SICEIA-2025-000778).

At both baseline and post-intervention, participants were scheduled in the morning following an overnight fast of 8-10 hours. They were instructed to maintain their usual lifestyle, abstain from alcohol and caffeine for 24 hours, and avoid strenuous physical activity for 72 hours prior to testing. Procedures included body composition assessment through electrical bioimpedance, a vastus lateralis muscle biopsy, fasting blood collection, and an oral glucose tolerance test (OGTT) by ingesting 75 grams of glucose and blood draws at 30, 60, 90, 120, 150, and 180 minutes post-ingestion. The same protocol was repeated after the 12-week intervention, with exercise groups completing their final training session at least 72 hours before the post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2D or prediabetes (glycated hemoglobin ≥ 5.7%)
* No history of substance abuse (tobacco, alcohol, or other drugs).
* Body mass index >25 kg/m², maintaining the habitual dietary patterns with stable body weight for at the least 6 months
* Stable physical activity and medication regimen for at least 6 months
* Not insulin-dependent
* Absence of injury, disease, disability, or other known medical condition which could affect the ability to successfully participate in physical exercise tests
* Absence of tumours and cancer disease
* Absence of other pathologies that could affect the study outcomes.
* Not under medication regimen that could affect the study outcomes.
* Being able to understand a communication in Spanish or English.
* Not pregnant

Exclusion Criteria:

* Failure to attend more than 2 consecutive or a total of 4 sessions of nutritional intervention.
* Failure to attend more than 4 consecutive or a total of 6 sessions of physical training.
* Serious injury
* Voluntary withdrawal
* Increased dose of diabetes medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle biopsy samples: mitochondrial respiratory capacity | Pre and post the 12-week intervention
  Skin was locally anesthetized, followed by an incision of approximately 6-7mm on the dermal surface. Using sterilized Bergstrom needles, approximately 3-6 mg of skeletal muscle from the lateral vastus were extracted and placed in a BIOPS buffer for immediate analysis of mitochondrial respiration (MR) through high-resolution respirometry. Before, the fibers were mechanically separated in BIOPS buffer using sterilized needles and chemically permeabilized with a 50 μg/ml saponin solution.
  MR was measured in a specific buffer (Mir05) in duplicate in hyperoxygenated chambers (250-450 mM of oxygen) in an Oxygraph-2k at 37ºC (Oroboros, Innsbruck, Austria). A substrate-uncoupler titration protocol was employed by adding (final concentration): malate (2mM), pyruvate (5mM), glutamate (2mM), MgCl2 (3mM), and ADP (5mM), cytochrome C (10μM), succinate (10mM), and p-trifluoromethoxyphenylhydrazone. Oxygen flux was presented as mass-specific (pmol·s/mg wet weight) and normalized to CS activity.
Assessed changes in Oxidative Stress | Pre and post the 12-week intervention
  The level of oxidative stress was assessed by the concentration of 8-OHdG as a biomarker of DNA oxidation. A competitive ELISA detection method was employed in serum samples. Briefly, the standard and the sample were added to a pre-coated microplate along with the biotinylated detection antibody. After washing, HRP-Streptavidin was added. Then, the TMB substrate was added, and the reaction was terminated with an acid solution. The color production was measured spectrophotometrically at a wavelength of 450nm. The optical density values of samples were compared with those of the standard curve to determine the 8-OHdG concentration (ng/ml).
Muscle biopsy sample: Citrate Synthase activity | Pre and post the 12-week intervention
  2-5 mg of frozen muscle was homogenized in a 1:20 dilution of CelLytic™ MT Tissue Lysis (C3228, Sigma-Aldrich, Dorset, UK), with 1 % protease inhibitor cocktail (P8340, Sigma-Aldrich, Dorset, UK) at 4 °C. The lysate was centrifuged at 12,000 × g for 10 min at 4 °C to pellet debris, and the supernatant was stored at -80 °C. CS activity was quantified in duplicates using an assay kit following the manufacturer's instructions (CS0720: Sigma-Aldrich, Dorset, UK). Briefly, endogenous activity was recorded through color emission by DTNB, and total activity was calculated after the addition of oxalacetate. Protein concentration was determined in duplicates using a bicinchoninic acid assay kit (BCA1: Sigma-Aldrich, Dorset, UK), enabling normalization of CS activity values to total protein content (µmol/g/min). CS activity and protein concentration were measured in 96-well plates using a microplate reader at 412 nm and 562 nm, respectively (MQX200R2, Biotek instruments, Burlington, USA).
Assessed changes in haemoglobin saturation delta | Pre and post the 12-week intervention
  A NIRO-200NX device was used to measure skeletal muscle changes on oxygenated, desoxygenated, and total haemoglobin (μmol/L) through near-infrared spectroscopy (NIRS) and the modified Beer-Lambert law. The NIRS sensor (emitter-sensor distance of 4cm) was placed at 2/3 of the distance between the major trochanter and the lateral epicondyle of the dominant leg. For parameters determined by MBLL, the reference point was set after five minutes of resting in a supine position. The NIRS data were continuously acquired throughout a resting energy expenditure test for 30 minutes, a maximal fat oxidation (MFO) test on a cycloergometer, and a maximal oxygen consumption (VO2max) test on a cycloergometer. Briefly, the MFO test consisted of an incremental task with 3-minute phases starting from 15W and increasing by 15W each phase until a respiratory exchange ratio of 1. After a 5-minute rest, the VO2max test was initiated at last MFO load with 15W increases each minute until VO2max determination.
Assessed changes in Tissue Oxygenation Index | Pre and post the 12-week intervention
  A NIRO-200NX device was used to measure skeletal muscle tissue oxygenation index (%)through near-infrared spectroscopy (NIRS), the modified Beer-Lambert law (MBLL), and spatially resolved spectroscopy. The NIRS sensor (emitter-sensor distance of 4cm) was placed at 2/3 of the distance between the major trochanter and the lateral epicondyle of the dominant leg. For parameters determined by MBLL, the reference point was set after five minutes of resting in a supine position. The NIRS data were continuously acquired throughout a resting energy expenditure test for 30 minutes, a maximal fat oxidation (MFO) test on a cycloergometer, and a maximal oxygen consumption (VO2max) test on a cycloergometer. Briefly, the MFO test consisted of an incremental task with 3-minute phases starting from 15W and increasing by 15W each phase until a respiratory exchange ratio of 1. After a 5-minute rest, the VO2max test was initiated at last MFO load with 15W increases each minute until VO2max determination.

SECONDARY OUTCOMES:
Assessed changes in Body composition: Fat mass and Fat-free mass. | Pre and post the 12-week intervention
  Body composition was estimated using a multifrequency bioimpedance of 8 electrodes previously validated (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) with at least 8 hours of fasting, and following these considerations the day before: 1) maintain their usual lifestyle, 2) refrain from consuming alcohol or caffeine for 24 hours, and 3) avoid vigorous physical activity for 72 hours before testing. Additionally, participants were asked to urinate just before the measurement.
  The patients wore light clothing and assumed a posture in accordance with the manufacturer's instructions.
  Additionally, body weight with the same device and height with a wall-mounted stadiometer (TANITA-LEICESTER HR-001, Tanita Corp., Tokyo, Japan) were measured in order to calculate body mass index.
Assessed changes in Glucose concentration | Pre and Post the 12-week intervention
  Glucose concentration (mg/dL) was measured from blood samples collected from the antecubital vein after at least 8 hours of fasting and at 30, 60, 90, 120, and 180 minutes after the ingestion of 75 grams of glucose (Nuter-tec, 75 g/200 mL, orange flavor). Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine consumption for 24 hours, and avoid vigorous physical activity for 72 hours. Blood samples were centrifuged at 4000 rpm for 7 minutes, and serum was analyzed. Glucose concentrations were determined using the colorimetric method performed on the Alinity CI system (Abbott Laboratories, Abbott Park, IL, USA).
Assessed changes in Insulin concentration | Pre and Post the 12-week intervention
  Insulin concentration (µU/mL) was measured from blood samples collected from the antecubital vein into serum separator tubes after at least 8 hours of fasting and at 30, 60, 90, 120, and 180 minutes after the ingestion of 75 grams of glucose (Nuter-tec, 75 g/200 mL, orange flavor). Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine consumption for 24 hours, and avoid vigorous physical activity for 72 hours. Blood samples were centrifuged at 4000 rpm for 7 minutes, and serum was analyzed. Insulin concentrations were determined by chemiluminescent immunoassays performed on the Alinity CI system (Abbott Laboratories, Abbott Park, IL, USA).
Assessed changes in Insulin Resistance: HOMA-IR | Pre and Post 12-week intervention
  Insulin resistance was estimated using the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), calculated as fasting insulin (µU/mL) multiplied by fasting glucose (mg/dL) divided by 405.
Assessed changes in Insulin Sensitivity: Matsuda Index | Pre and Post 12-week intervention
  Whole body insulin sensitivity was estimated through the Matsuda Index, calculated as 10,000 / √[(fasting glucose (mg/dL) × fasting insulin (µU/mL)) × (mean glucose during Oral Glucose Tolerance Test (mg/dL) × mean insulin during Oral Glucose Tolerance Test (µU/mL))].
Assessed changes in Insulin Sensitivity: Quicki | Pre and Post 12-week intervention
  Insulin sensitivity was estimated through the Quantitative Insulin Sensitivity Check Index (QUICKI), calculated as 1 / [log(fasting insulin (µU/mL)) + log(fasting glucose (mg/dL))].
Assessed changes in Body Weight | Pre and Post the 12-week intervention
  Body weight (kilograms, kg) was measured using a multifrequency bioelectrical impedance device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed Height | Pre and Post 12-week Intervention
  Height (meters, m) was measured using a wall-mounted stadiometer (TANITA-LEICESTER HR-001, Tanita Corp., Tokyo, Japan) with participants standing in accordance with the manufacturer's instructions.
Assessed changes in Body Mass Index | Pre and Post 12-week Intervention
  Body Mass Index (BMI) in kilograms per square meter (kg/m²) was calculated as body weight (kg) divided by height squared (m²).
Assessed changes in Fat Mass (kilograms of Fat Mass) | Pre and Post 12-week Intervention
  Fat mass (kilograms, kg) was estimated using multifrequency bioelectrical impedance with an 8-electrode device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed changes in Fat Mass (percentage of Fat Mass) | Pre and Post 12-week Intervention
  Fat mass (percentage of total body weight, %) was estimated using multifrequency bioelectrical impedance with an 8-electrode device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed changes in Fat-free Mass (kilograms of Fat-free Mass) | Pre and Post 12-week Intervention
  Fat-free mass (kilograms, kg) was estimated using multifrequency bioelectrical impedance with an 8-electrode device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed changes in Fat-free Mass (percentage of Fat-free Mass) | Pre and Post 12-week Intervention
  Fat-free mass (percentage of total body weight, %) was estimated using multifrequency bioelectrical impedance with an 8-electrode device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed changes in Anthropometry: Perimeters | Pre and Post 12-week Intervention
  Waist circumference (cm) was measured at the midpoint between the lower lateral margin of the 10th rib and the iliac crest, perpendicular to the longitudinal axis of the trunk. Abdominal circumference (cm) was measured at the level of the umbilicus, perpendicular to the longitudinal axis of the trunk. Hip circumference (cm) was measured at the level of the greatest posterior prominence of the buttocks, perpendicular to the longitudinal axis of the trunk. Thigh circumference (cm) was measured at the midpoint between the greater trochanter and the lateral tibial condyle. All measurements were performed with the participant standing upright, and relaxed. Each measurement was taken twice, and a third measurement was performed if the difference exceeded 1%. The mean of the two most similar records was registered.
Assessed changes in Anthropometry: Waist to Hip Ratio | Pre and Post 12-week Intervention
  Waist-to-hip ratio (WHR) was calculated as waist circumference (cm) divided by hip circumference (cm).
Assessed changes in Anthropometry: Skinfold thickness | Pre and Post 12-week Intervention
  Thigh skinfold thickness was measured at two-thirds of the distance from the iliospinale point (the lowest part of the anterior superior iliac spine) to the superolateral border of the patella, over the belly of the vastus lateralis muscle. Measurements were taken on the dominant leg. Two measurements were obtained, and a third was taken if the difference between the first two exceeded 5%. The mean of the two most similar records was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Casals Vázquez, PhD, Principal Investigator — University of Cádiz; Miguel Efrén Jiménez Romero, MD, Principal Investigator — Hospital de la Línea de la Concepción
Locations (1):
- Science of Education Faculty, Puerto Real, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: No